CLINICAL TRIAL: NCT01695499
Title: Open, Prospective, Multicenter Trial to Evaluate the Clinical Significance of Combined Serological (Galactomannan ELISA, Beta D Glucan Assay) and Molecular (Nested Aspergillus PCR Assay, Real-time qPCR Assay, Multifungal DNA Microarray) Diagnostic Assays to Detect and Characterize Fungal Pathogens in Bronchoalveolar Lavage (BAL)and Blood Samples of Intensive Care Unit Patients With Pulmonary Infiltrates
Brief Title: Diagnostic Study of Biomarkers in BAL of ICU Patients With Lung Infiltrates
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heidelberg University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dieter Buchheidt, Professor Dr. Dieter Buchheidt, Heidelberg University
Other Study IDs: BAL-Biomarker-ICU Study; Grant Pfizer ASPIRE Award (Other Grant/Funding Number: Pfizer Grant # WS 2274964)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: INvasive Aspergillosis; Mechanical Ventilation; Lung Infiltrates; Diagnostics; Biomarker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Only fungal DNA investigated
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Immunosuppressed ICU Patients with lung infiltrates: Immunosuppressed ICU Patients with lung infiltrates
- Control Group: BAL and blood aliquots of 20 immunocompetent pts (suffering from lung diseases) will be collected and tested identically as a control population.

SUMMARY:
The aim of this project is therefore to explore on the clinical significance of analyzing surrogate markers combined with conventional diagnostics in the ICU setting. BAL, blood and biopsy samples will be subjected to a combined analysis of GM, BDG, Aspergillus specific PCR assays in addition to conventional diagnostics (Microscopy, Culture,Histology) for ICU pts with pulmonary infiltrates.

As GM and BDG are not species-specific, three established and repeatedly published species specific PCR-based assays (nested PCR, real time PCR assay, multifungal DNA Array)developed by our group will be investigated in combination with the serological tests in a multicenter prospective clinical diagnostic trial.

ELIGIBILITY:
Inclusion Criteria:

* underlying conditions (see above)
* being on mechanical ventilation
* lung infiltrates

Exclusion Criteria:

* immunocompetent patients (not fulfilling the criteria above)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Immunocompromised patients on the intensive care unit with lun infiltrates and one of the following underlying conditions:
  * Underlying malignancy
  * Antineoplastic chemotherapy
  * Neutropenia
  * Allogeneic hematopoietic stem cell transplantation
  * Solid organ transplantation
  * Retransplantation
  * Acute or chronic immunological rejection or graft-versus-host-disease
  * Treatment with immunosuppressive agents (calcineurin inhibitors, OKT3, etc)
  * Profound systemic corticosteroid therapy prior to ICU admission
  * COPD Gold III/IV
  * Advanced liver cirrhosis and ICU treatment for more than 7 days
  * Hemodialysis, renal failure
  * CMV infection
  * HIV infection; CD4 cellcount
  * Post splenectomy
  * Post cardiac surgery
  * Diabetes mellitus
  * mechanical ventilation for more than 21 days
  * ICU-based steroid therapy and corticosteroid treatment for more than 7 days
  * Malnutrition
  * Severe burn wounds
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of combined biomarker testing in BAL fluid in relation to diagnostic certainty | 6 weeks
  Evaluation of diagnostic accuracy of the combined biomarker approach

CONTACTS AND LOCATIONS:
Locations (1):
- Mannheim University Hospital, Mannheim, Germany

REFERENCES:
- [Background] Reinwald M, Hummel M, Kovalevskaya E, Spiess B, Heinz WJ, Vehreschild JJ, Schultheis B, Krause SW, Claus B, Suedhoff T, Schwerdtfeger R, Reuter S, Kiehl MG, Hofmann WK, Buchheidt D. Therapy with antifungals decreases the diagnostic performance of PCR for diagnosing invasive aspergillosis in bronchoalveolar lavage samples of patients with haematological malignancies. J Antimicrob Chemother. 2012 Sep;67(9):2260-7. doi: 10.1093/jac/dks208. Epub 2012 Jun 27. PMID 22740590
- [Background] Reinwald M, Spiess B, Heinz WJ, Vehreschild JJ, Lass-Florl C, Kiehl M, Schultheis B, Krause SW, Wolf HH, Bertz H, Maschmeyer G, Hofmann WK, Buchheidt D. Diagnosing pulmonary aspergillosis in patients with hematological malignancies: a multicenter prospective evaluation of an Aspergillus PCR assay and a galactomannan ELISA in bronchoalveolar lavage samples. Eur J Haematol. 2012 Aug;89(2):120-7. doi: 10.1111/j.1600-0609.2012.01806.x. Epub 2012 Jun 22. PMID 22650156
- [Background] Spiess B, Seifarth W, Merker N, Howard SJ, Reinwald M, Dietz A, Hofmann WK, Buchheidt D. Development of novel PCR assays to detect azole resistance-mediating mutations of the Aspergillus fumigatus cyp51A gene in primary clinical samples from neutropenic patients. Antimicrob Agents Chemother. 2012 Jul;56(7):3905-10. doi: 10.1128/AAC.05902-11. Epub 2012 Apr 23. PMID 22526309
- [Derived] Boch T, Reinwald M, Spiess B, Liebregts T, Schellongowski P, Meybohm P, Rath PM, Steinmann J, Trinkmann F, Britsch S, Michels JD, Jabbour C, Hofmann WK, Buchheidt D. Detection of invasive pulmonary aspergillosis in critically ill patients by combined use of conventional culture, galactomannan, 1-3-beta-D-glucan and Aspergillus specific nested polymerase chain reaction in a prospective pilot study. J Crit Care. 2018 Oct;47:198-203. doi: 10.1016/j.jcrc.2018.07.001. Epub 2018 Jul 4. PMID 30015290